CLINICAL TRIAL: NCT02648477
Title: MK-3475 (Pembrolizumab) in Combination With an Anthracycline or Anti-estrogen Therapy in Patients With Triple Negative and Hormone Receptor Positive (HR+ HER2-) Metastatic Breast Cancer
Brief Title: Pembrolizumab and Doxorubicin Hydrochloride or Anti-Estrogen Therapy in Treating Patients With Triple-Negative or Hormone Receptor-Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15295; NCI-2015-02194 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15295 (Other: City of Hope Medical Center)
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Results first posted 2023-04-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Estrogen Receptor Negative; Estrogen Receptor Positive; HER2/Neu Negative; Progesterone Receptor Negative; Progesterone Receptor Positive; Stage IV Breast Cancer; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Anastrozole; Doxorubicin; exemestane; Letrozole; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (pembrolizumab, doxorubicin hydrochloride) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 and doxorubicin hydrochloride IV on day 1. Treatment repeats every 3 weeks for 6 courses, and then continues for up to 24 months with pembrolizumab alone in the absence of disease progression or unacceptable toxicity.
  Patients who stop pembrolizumab with stable disease or better may receive additional pembrolizumab therapy for up to 1 year if they progress after stopping study treatment.
  Interventions: Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab
- Cohort 2 (pembrolizumab, anti-estrogen therapy) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 and an aromatase inhibitor (exemestane, anastrozole, or letrozole) PO QD on days 1-21. Treatment repeats every 3 weeks for 24 months in the absence of disease progression or unacceptable toxicity.
  In both arms, patients who stop pembrolizumab with stable disease or better may receive additional pembrolizumab therapy for up to 1 year if they progress after stopping study treatment.
  Interventions: Drug: Anastrozole; Drug: Exemestane; Other: Laboratory Biomarker Analysis; Drug: Letrozole; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Anastrozole — Given PO
  Other Names: Arimidex; ICI D1033; ICI-D1033; ZD-1033
  Arms: Cohort 2 (pembrolizumab, anti-estrogen therapy)
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
  Arms: Cohort 1 (pembrolizumab, doxorubicin hydrochloride)
Drug: Exemestane — Given PO
  Other Names: Aromasin; FCE-24304
  Arms: Cohort 2 (pembrolizumab, anti-estrogen therapy)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Letrozole — Given PO
  Other Names: CGS 20267; Femara
  Arms: Cohort 2 (pembrolizumab, anti-estrogen therapy)
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab and doxorubicin hydrochloride works compared to pembrolizumab with anti-estrogen therapy (anastrozole, letrozole, or exemestane) in treating patients with triple-negative or hormone-receptor positive breast cancer that has spread from the primary site (place where it started) to other places in the body. Pembrolizumab is an antibody drug that blocks a molecule called programmed death (PD)-1. PD-1 is a molecule that shuts down the body's immune responses and prevents the immune system from attacking the cancer. Doxorubicin hydrochloride is a drug used in chemotherapy that works to stop the growth of tumor cells by stopping them from dividing and by causing them to die. Anti-estrogen therapy, including anastrozole, letrozole, and exemestane, lowers estrogen levels in the body, which may help treat cancer that is hormone receptor-positive. Giving pembrolizumab together with standard treatment of either doxorubicin hydrochloride (triple-negative cancer) or anti-estrogen therapy (hormone receptor-positive cancer) may be an effective treatment for these types of breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate efficacy (overall response rate) of MK-3475 (pembrolizumab) and doxorubicin (doxorubicin hydrochloride) in patients with stage IV triple negative breast cancer.

II. To evaluate efficacy (overall response rate) of MK-3475 and an oral aromatase inhibitor in patients with stage IV hormone receptor positive (HR+) human epidermal growth factor receptor 2 negative (HER2-) breast cancer.

SECONDARY OBJECTIVES:

I. To assess clinical benefit rate (lack of progression for > 24 weeks), duration of response, time-to-treatment failure, progression-free survival, and overall survival in triple negative (TN) stage IV breast cancer patients based primarily on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and immune-related (ir)RECIST.

II. To assess feasibility and toxicity.

III. To assess clinical benefit rate (lack of progression for > 24 weeks), duration of response, time-to-treatment failure, progression-free survival, and overall survival in patients with stage IV HR+ breast cancer based primarily on RECIST 1.1, and irRECIST.

IV. To assess feasibility and toxicities.

TERTIARY OBJECTIVES:

I. To procure serial tumor (primary and metastatic) and blood (cellular and serum/plasma) samples and analyze them to better our understanding of cellular and humoral immune response correlates and predictors of clinical benefits, leading to optimized selection of target populations in future phase II and subsequent phase III randomized prospective trials.

OUTLINE: Patients are assigned to 1 of 2 treatment arms.

COHORT 1 (TRIPLE-NEGATIVE): Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 and doxorubicin hydrochloride IV on day 1. Treatment repeats every 3 weeks for 6 courses, and then continues for up to 24 months with pembrolizumab alone in the absence of disease progression or unacceptable toxicity.

COHORT 2 (HORMONE/HER2+): Patients receive pembrolizumab IV over 30 minutes on day 1 and an aromatase inhibitor (exemestane, anastrozole, or letrozole) orally (PO) once daily (QD) on days 1-21. Treatment repeats every 3 weeks for 24 months in the absence of disease progression or unacceptable toxicity.

In both arms, patients who stop pembrolizumab with stable disease or better may receive additional pembrolizumab therapy for up to 1 year if they progress after stopping study treatment.

After completion of study treatment, patients are followed up for 30 days after the end of treatment and then every 8-12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 1) stage IV metastatic triple negative breast cancer (triple negative is defined as estrogen receptor [ER] and progesterone receptor [PgR] status is < 1% of tumor cell nuclei are immunoreactive for ER or PgR, and HER2 status is fluorescence in situ hybridization [FISH] negative or immunohistochemistry [IHC] 0 or 1+), or 2) stage IV HR+ HER2- (HR+) breast cancer (defined as ER or PgR > 1% of tumor cell nuclei are immunoreactive for ER or PgR and HER2 statis is FISH negative or IHC - or 1+)
* Be willing and able to provide written informed consent/assent for the trial
* Have measurable disease based on RECIST 1.1
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion; newly-obtained in defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on day 1; subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the sponsor
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Serum creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance >= 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]); creatinine clearance should be calculated per institutional standard
* Left ventricular ejection fraction by multigated acquisition scan (MUGA) or echocardiogram >= 55% for patients with triple negative breast cancer; >= upper limit of institutional normal for patient with HR+ breast cancer
* Serum total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN OR =< 5 x ULN for subjects with liver metastases
* Albumin >= 2.5 mg/dL
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Reproductive status for cohort 2: HR+ stage IV post-menopausal breast cancer; post-menopausal is defined by at least one of the following criteria:

  * Prior bilateral oophorectomy OR amenorrheic for >= 12 months (if =< 55 years of age and prior chemotherapy or on medical ovarian ablative therapy or received ovarian radiation for ablation in the past 5 years and/or tamoxifen or an aromatase inhibitor (AI) within the past year, then follicle-stimulating hormone (FSH) and estradiol must be in the post-menopausal range and obtained within 28 days prior to registration) OR
  * Previous hysterectomy with one or both ovaries left in place (or previous hysterectomy in which documentation of bilateral oophorectomy is unavailable AND FSH values consistent with the institutional normal values for the post-menopausal state; FSH levels must be obtained within 28 days prior to registration
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Subjects currently on a bisphosphonate or denosumab are eligible for study therapy

Exclusion Criteria:

* Cohort 1: Has triple negative breast cancer, is considered for cohort 1 participation, and received prior anthracycline therapy
* Cohort 2: Has received prior aromatase inhibitor therapy and is deemed to be resistant to all three (anastrozole, letrozole, exemestane) approved AIs; resistance is defined as progression within 12 months or while on an AI
* Patient is premenopausal (medical ovarian suppression is allowed); is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active TB (Bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Suboptimal cardiac function as defined by decreased left ventricular ejection fraction < 55% for cohort 1, and < 50% for cohort 2
* Prior pembrolizumab
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent; Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study; Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that has progressed or required active treatment in the past 5 years; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of, active pneumonitis requiring treatment with steroids or history of/active interstitial lung disease
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-programmed death-ligand (PD-L)1, or anti-PD-L2 agent
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has a history of (non-infectious) pneumonitis that required steroids or currently has pneumonitis
* Has received a live vaccine within 30 days of planned start of study therapy; Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Waisman, MD, Principal Investigator — City of Hope Medical Center
Locations (6):
- United States (6):
  - City of Hope Corona, Corona, California
  - City of Hope Medical Center, Duarte, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope Rancho Cucamonga, Rancho Cucamonga, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope West Covina, West Covina, California

REFERENCES:
- [Derived] Egelston CA, Guo W, Yost SE, Ge X, Lee JS, Frankel PH, Cui Y, Ruel C, Schmolze D, Murga M, Tang A, Martinez N, Karimi M, Somlo G, Lee PP, Waisman JR, Yuan Y. Immunogenicity and efficacy of pembrolizumab and doxorubicin in a phase I trial for patients with metastatic triple-negative breast cancer. Cancer Immunol Immunother. 2023 Sep;72(9):3013-3027. doi: 10.1007/s00262-023-03470-y. Epub 2023 Jun 9. PMID 37294342

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (Pembrolizumab, Doxorubicin Hydrochloride) Triple Negative Breast Cancer: Pembrolizumab 200 mg IV every 3 weeks and doxorubicin 50-60 mg/m2 IV every 3 weeks x 6 cycles followed by a pembrolizumab alone for up to 35 cycles or a maximum of 24 months starting from the first cycle.
  Patients who stop pembrolizumab with stable disease or better may receive additional pembrolizumab therapy for up to 1 year if they progress after stopping study treatment.
  Doxorubicin Hydrochloride: Given IV
  Pembrolizumab: Given IV
- Cohort 2 (Pembrolizumab, Anti-estrogen Therapy) HR+ HER2- Breast Cancer: Pembrolizumab 200 mg IV every 3 weeks and anastrozole 1 mg, letrozole 2.5 mg, or exemestane 25 mg (preferred) daily.
  Treatment repeats every 3 weeks for 24 months in the absence of disease progression or unacceptable toxicity.
  Patients who stop pembrolizumab with stable disease or better may receive additional pembrolizumab therapy for up to 1 year if they progress after stopping study treatment.
  Anastrozole: Given PO
  Exemestane: Given PO
  Letrozole: Given PO
  Pembrolizumab: Given IV
Period: Overall Study
Arm/Group | Cohort 1 (Pembrolizumab, Doxorubicin Hydrochloride) Triple Negative Breast Cancer | Cohort 2 (Pembrolizumab, Anti-estrogen Therapy) HR+ HER2- Breast Cancer
Started | 10 | 20
Completed | 10 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Pembrolizumab, Doxorubicin Hydrochloride) Triple Negative Breast Cancer | Cohort 2 (Pembrolizumab, Anti-estrogen Therapy) HR+ HER2- Breast Cancer | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Continuous [Median (Full Range); unit: years] | 62 [41 to 87] | 62 [34 to 79] | 62 [34 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 20 | 30
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 3 | 5
  White | 7 | 15 | 22
  Pacific Islander | 0 | 1 | 1
  Unknown | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 20 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Pembrolizumab, Doxorubicin Hydrochloride) Triple Negative Breast Cancer | Cohort 2 (Pembrolizumab, Anti-estrogen Therapy) HR+ HER2- Breast Cancer
Number analyzed (Participants) | 10 | 20
Participants | 5 | 2

2. Secondary Outcome: Clinical Benefit Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI:
  Complete Response (CR), Disappearance of all target lesions; Partial response (PR): At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR; Stable disease (SD): Neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD; Progressive disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). Clinical Benefit Rate (CBR) = CR + PR + SD at 6 months
Time Frame: Up to 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (Pembrolizumab, Doxorubicin Hydrochloride) Triple Negative Breast Cancer | Cohort 2 (Pembrolizumab, Anti-estrogen Therapy) HR+ HER2- Breast Cancer
Number analyzed (Participants) | 10 | 20
percentage of participants | 50 | 20

3. Secondary Outcome: Overall Survival (OS)
Description: Estimated using the product-limit method of Kaplan and Meier. From initial treatment until death from any cause.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (Pembrolizumab, Doxorubicin Hydrochloride) Triple Negative Breast Cancer | Cohort 2 (Pembrolizumab, Anti-estrogen Therapy) HR+ HER2- Breast Cancer
Number analyzed (Participants) | 10 | 20
Months | 15.6 [13.3 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 17.2 [9.4 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Estimated using the product-limit method of Kaplan and Meier. Failure defined as disease progression or death from any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (Pembrolizumab, Doxorubicin Hydrochloride) Triple Negative Breast Cancer | Cohort 2 (Pembrolizumab, Anti-estrogen Therapy) HR+ HER2- Breast Cancer
Number analyzed (Participants) | 10 | 20
Months | 5.2 [4.7 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 1.8 [1.6 to 2.6]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time of initial treatment until 30 days post discontinuation of treatment, up to 3 years.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Cohort 1 (Pembrolizumab, Doxorubicin Hydrochloride) Triple Negative Breast Cancer | Cohort 2 (Pembrolizumab, Anti-estrogen Therapy) HR+ HER2- Breast Cancer
All-Cause Mortality (participants affected / at risk) | 7/10 | 16/20
Serious Adverse Events (participants affected / at risk) | 3/10 | 2/20
Other Adverse Events (participants affected / at risk) | 10/10 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Pembrolizumab, Doxorubicin Hydrochloride) Triple Negative Breast Cancer (N=10) | Cohort 2 (Pembrolizumab, Anti-estrogen Therapy) HR+ HER2- Breast Cancer (N=20)
Heart failure (Cardiac disorders) | 1 (2) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, spe (Infections and infestations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Pembrolizumab, Doxorubicin Hydrochloride) Triple Negative Breast Cancer (N=10) | Cohort 2 (Pembrolizumab, Anti-estrogen Therapy) HR+ HER2- Breast Cancer (N=20)
Anemia (Blood and lymphatic system disorders) | 8 (23) | 7 (12)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (2) | 1 (2)
Palpitations (Cardiac disorders) | 1 (1) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 3 (5) | 0 (0)
Ear and labyrinth disorders - Other, spe (Ear and labyrinth disorders) | 1 (6) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (2)
Blurred vision (Eye disorders) | 0 (0) | 1 (4)
Conjunctivitis (Eye disorders) | 2 (3) | 0 (0)
Dry eye (Eye disorders) | 2 (3) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 7 (11)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (4) | 3 (5)
Constipation (Gastrointestinal disorders) | 4 (5) | 6 (20)
Diarrhea (Gastrointestinal disorders) | 4 (10) | 5 (9)
Dry mouth (Gastrointestinal disorders) | 2 (3) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (4) | 2 (3)
Gastrointestinal disorders - Other, spec (Gastrointestinal disorders) | 0 (0) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 3 (9) | 3 (3)
Nausea (Gastrointestinal disorders) | 9 (36) | 7 (12)
Oral pain (Gastrointestinal disorders) | 1 (3) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (11) | 1 (1)
Chills (General disorders) | 4 (4) | 2 (3)
Edema limbs (General disorders) | 2 (4) | 4 (4)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 9 (49) | 15 (59)
Fever (General disorders) | 1 (1) | 1 (2)
Flu like symptoms (General disorders) | 1 (3) | 1 (11)
General disorders and administration sit (General disorders) | 3 (4) | 1 (15)
Localized edema (General disorders) | 3 (4) | 3 (4)
Malaise (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2) | 1 (1)
Pain (General disorders) | 5 (6) | 3 (4)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, spe (Infections and infestations) | 1 (2) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (4) | 1 (4)
Alanine aminotransferase increased (Investigations) | 2 (4) | 8 (32)
Alkaline phosphatase increased (Investigations) | 0 (0) | 10 (27)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 9 (29)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (8)
Creatinine increased (Investigations) | 2 (5) | 2 (37)
Electrocardiogram QT corrected interval (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 6 (20) | 2 (5)
Neutrophil count decreased (Investigations) | 6 (15) | 0 (0)
Platelet count decreased (Investigations) | 2 (5) | 5 (7)
Weight gain (Investigations) | 0 (0) | 1 (2)
Weight loss (Investigations) | 3 (9) | 3 (4)
White blood cell decreased (Investigations) | 9 (28) | 7 (20)
Acidosis (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 5 (9) | 6 (23)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2) | 6 (11)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (4) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (3) | 3 (5)
Hypokalemia (Metabolism and nutrition disorders) | 6 (14) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 5 (11) | 7 (14)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 4 (6)
Metabolism and nutrition disorders - Oth (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (23)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (9) | 7 (43)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (7)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (4) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (5)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Musculoskeletal and connective tissue di (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (22)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (10)
Neoplasms benign, malignant and unspecif (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 2 (9)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (12)
Headache (Nervous system disorders) | 3 (6) | 5 (15)
Memory impairment (Nervous system disorders) | 2 (7) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (16) | 4 (13)
Phantom pain (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 2 (9)
Anxiety (Psychiatric disorders) | 4 (5) | 3 (24)
Depression (Psychiatric disorders) | 1 (1) | 6 (26)
Insomnia (Psychiatric disorders) | 2 (10) | 7 (37)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 4 (10) | 0 (0)
Proteinuria (Renal and urinary disorders) | 4 (7) | 2 (2)
Renal and urinary disorders - Other, spe (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 2 (3)
Urinary tract pain (Renal and urinary disorders) | 1 (2) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (8)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 5 (17)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (8)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal di (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (6) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (4) | 3 (11)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (7) | 5 (12)
Flushing (Vascular disorders) | 1 (1) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 7 (37)
Hypertension (Vascular disorders) | 8 (47) | 7 (59)
Hypotension (Vascular disorders) | 1 (1) | 3 (4)
Thromboembolic event (Vascular disorders) | 1 (2) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT02648477/Prot_SAP_000.pdf